CLINICAL TRIAL: NCT02564718
Title: 7-day Study of the Safety, Efficacy and the Pharmacokinetic and Pharmacodynamic Properties of Oral Rivaroxaban in Children From Birth to Less Than 6 Months With Arterial or Venous Thrombosis
Brief Title: Rivaroxaban for Treatment in Venous or Arterial Thrombosis in Neonates
Acronym: Einstein Jr
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17618; 2014-002385-74 (EudraCT Number)
Record Dates: First submitted 2015-09-04; First posted 2015-10-01 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Thromboembolism
Keywords: Pediatric
MeSH Terms: conditions — Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Rivaroxaban oral suspension from granules will be dosed according to body weight as oral 0.1% suspension (1 mg/mL)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Body weight adjusted dosing of rivaroxaban to achieve a similar exposure in the range as that observed in adults treated for venous thromboembolism (VTE) with 20 mg once daily.

SUMMARY:
The purpose of this study is to find out whether rivaroxaban is safe and effective to use in children age newborn to less than 6 months and how long it stays in the body and how it is used in the body. Safety will be assessed by looking at the incidence and types of bleeding events. There will also be a check for worsening of blood clots.

DETAILED DESCRIPTION:
Neonates and infants aged less than 6 months who pass the screen of in- and exclusion criteria, who have been treated for at least five days with heparin and /or vitamin K antagonist (VKA) for confirmed symptomatic or asymptomatic arterial or venous thrombosis are eligible for the study. Study treatment consists of a 7-day treatment with an age- and body weight-adjusted three times daily, approximately 8 hours apart oral rivaroxaban dosing to achieve a similar exposure as that observed in adults treated for venous thromboembolism (VTE) with 20 mg rivaroxaban once daily. Rivaroxaban will be provided as granules for preparation of an oral suspension (1 mg/mL after re-suspension) using a t.i.d. regimen with 8-hour intervals. An ultrasound will be performed before starting rivaroxaban at treatment day 1 and after the end of rivaroxaban treatment at day 8. The last dose of rivaroxaban treatment will be followed by a 30-day post study treatment period, regardless of the duration of study drug administration. After cessation of rivaroxaban, it is at the investigator's discretion to continue with anticoagulants. The principal safety outcome is the combination of major and clinically relevant non-major bleeding. The efficacy outcome is the composite of all symptomatic recurrent thromboembolism and asymptomatic deterioration in thrombotic burden on repeat imaging. All suspected recurrent thromboembolism, asymptomatic deterioration in thrombotic burden on repeat imaging, deaths, as well as all episodes of bleeding will be evaluated by a central independent adjudication committee (CIAC). Adjudication results will be the basis for the final analyses.

For all children, visits are scheduled at regular time points (see Table 1). Enrolled children who are not treated or those with premature discontinuation of rivaroxaban will at least be seen at the end of the study treatment period. During all contacts, the treatment and clinical course of the child will be evaluated. Children with suspected efficacy or safety outcomes will undergo confirmatory testing as per standard of care. Blood samples for pharmacokinetic (PK)/pharmacodynamics (PD) will be taken at defined time points (see Table 2).

An Independent Data Monitoring Committee (DMC) will monitor the children's safety during the study and give recommendations to the steering committee.

ELIGIBILITY:
Inclusion Criteria:

* Children from birth to less than 6 months with documented symptomatic or asymptomatic venous or arterial thrombosis who have been treated with anticoagulant therapy for at least 5 days.
* Gestational age at birth of at least 37 weeks.
* Hemoglobin, platelets, creatinine, ALT and total and direct bilirubin assessed within 10 days prior to enrollment.
* Oral feeding/nasogastric/gastric feeding for at least 10 days.
* Informed consent provided.
* Body weight >2600 g

Exclusion Criteria:

* Active bleeding or high risk for bleeding contraindicating anticoagulant therapy, including history of intra-ventricular bleeding.
* Symptomatic progression of thrombosis during preceding anticoagulant treatment.
* Planned invasive procedures, including lumbar puncture and removal of non-peripherally placed central lines during study treatment.
* Hepatic disease which is associated with either: coagulopathy leading to a clinically relevant bleeding risk, or alanine aminotransferase (ALT) > 5x upper level of normal (ULN) or total bilirubin (TB) > 2x ULN with direct bilirubin > 20% of the total.
* Creatinine >1.5 times of normal.
* Uncontrolled Hypertension defined as >95th percentile.
* History of gastrointestinal disease or surgery associated with impaired absorption.
* Platelet count <100 x 109/L.
* Concomitant use of strong inhibitors of both cytochrome P450 isoenzyme 3A4 (CYP3A4) and P-glycoprotein (P-gp), e.g. all human immunodeficiency virus protease inhibitors and the following azole-antimycotics agents: ketoconazole, itraconazole, voriconazole, posaconazole, if used systemically (fluconazole is allowed)
* Concomitant use of strong inducers of CYP3A4, e.g. rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
* Indication for anticoagulant therapy other than current thrombosis.
* Indication for antiplatelet therapy or non-steroid anti-inflammatory drug (NSAID) therapy. Incidental use is allowed.
* Hypersensitivity to rivaroxaban or its excipients.
* Participation in a study with an investigational drug or medical device within 30 days prior to enrollment.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Vienna, Austria
- Montpellier, France
- Erlangen, Germany
- Ramat Gan, Israel
- Milan, Lombardy, Italy
- Spain (2):
  - Barcelona
  - Madrid
- Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Monagle P, Lensing AWA, Thelen K, Martinelli I, Male C, Santamaria A, Samochatova E, Kumar R, Holzhauer S, Saracco P, Simioni P, Robertson J, Grangl G, Halton J, Connor P, Young G, Molinari AC, Nowak-Gottl U, Kenet G, Kapsa S, Willmann S, Pap AF, Becka M, Twomey T, Beyer-Westendorf J, Prins MH, Kubitza D; EINSTEIN-Jr Phase 2 Investigators. Bodyweight-adjusted rivaroxaban for children with venous thromboembolism (EINSTEIN-Jr): results from three multicentre, single-arm, phase 2 studies. Lancet Haematol. 2019 Oct;6(10):e500-e509. doi: 10.1016/S2352-3026(19)30161-9. Epub 2019 Aug 13. PMID 31420317
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 9 study centers in 7 countries between 19 November 2015 (first participant first visit) and 18 December 2017 (last participant last visit).
Pre-assignment Details: Overall, 11 participants were screened, of these 1 participant was not included in the study due to withdrawal by parent. A total of 10 participants were assigned to treatment.
Groups:
- Rivaroxaban (BAY59-7939) Suspension Bid: Participants aged less than 6 months were administered with age- and body weight-adjusted 0.5 to 3.2 milligram (mg) oral dose of rivaroxaban oral suspension twice daily (bid) for 7 days.
- Rivaroxaban (BAY59-7939) Suspension Tid: Participants aged less than 6 months were administered with age- and body weight-adjusted 0.5 to 2.9 mg oral dose of rivaroxaban oral suspension thrice daily (tid) for 7 days.
Period: Overall Study
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Withdrew from treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants who received at least one dose of rivaroxaban.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: SAF included all participants who received at least one dose of rivaroxaban.
  Months | 1.81 (2.24) | 1.12 (0.60) | 1.47 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: SAF included all participants who received at least one dose of rivaroxaban.
  Participants
    Female | 1 | 4 | 5
    Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: SAF included all participants who received at least one dose of rivaroxaban.
  Participants
    Black or African American | 1 | 0 | 1
    White | 3 | 5 | 8
    Unknown or Not Reported | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] — Population: SAF included all participants who received at least one dose of rivaroxaban.
  Kilogram (kg) | 4.33 (2.19) | 3.70 (0.85) | 4.02 (1.60)
Prothrombin Time [Mean (Standard Deviation); unit: Seconds (sec)] — Population: PD analysis set (PDS) included all participants with at least one blood sample for clotting parameters in accordance with the PD sampling strategy.
  Seconds (sec)
    number analyzed (Participants) | 5 | 4 | 9
    (all) | 13.3 (0.378) | 13.9 (1.31) | NA (NA) — Mean and Standard Deviation of Prothrombin Time values for the overall participants was not calculated.
Activated Partial Thromboplastin Time (aPTT) [Mean (Standard Deviation); unit: Seconds (sec)] — Population: PDS included all participants with at least one blood sample for clotting parameters in accordance with the PD sampling strategy.
  Seconds (sec)
    number analyzed (Participants) | 5 | 4 | 9
    (all) | 34.0 (4.05) | 34.9 (2.62) | NA (NA) — Mean and Standard Deviation of aPTT values for the overall participants was not calculated.

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Rivaroxaban in Plasma as a Measure of Pharmacokinetics at Day 1
Description: Concentration of pharmacokinetic parameters of rivaroxaban in plasma was evaluated.
Time Frame: 30 minutes to 1.5 hours post-dose; 2 to 4 hours post-dose (bid dosing) and 30 minutes to 3 hours post-dose; 7 to 8 hours post-dose on Day 1 (tid dosing)
Population: Pharmacokinetic (PK) analysis set (PKS) included all participants with at least one PK sample in accordance with the PK sampling strategy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L)
  30 minutes to 1.5 hours post-dose: number analyzed (Participants) | 5 | 0
  30 minutes to 1.5 hours post-dose | 85.2001 (37.72) |
  30 minutes to 3 hours post-dose: number analyzed (Participants) | 0 | 5
  30 minutes to 3 hours post-dose |  | 42.6837 (39.35)
  2 to 4 hours post-dose: number analyzed (Participants) | 5 | 0
  2 to 4 hours post-dose | 73.7641 (64.38) |
  7 to 8 hours post-dose: number analyzed (Participants) | 0 | 5
  7 to 8 hours post-dose |  | 12.1027 (130.13)

2. Secondary Outcome: Number of Participants With Major and Clinically Relevant Non-Major Bleeding Events
Description: Central independent adjudication committee (CIAC) classified bleeding as follows: Major bleeding is defined as overt bleeding and •associated with a fall in hemoglobin of 2 gram/deciliter (g/dL) or more, •leading to a transfusion of the equivalent of 2 or more units of packed red blood cells or whole blood in adults, or •occurring in a critical site, example: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal, or •contributing to death. Clinically relevant non-major bleeding is defined as overt bleeding not meeting the criteria for major bleeding, but associated with: •medical intervention, or •unscheduled contact (visit or telephone call) with a physician, or •cessation (temporary) of study treatment, or •discomfort for the child such as pain
Time Frame: From start of study drug administration until 30-day post study treatment period
Population: Safety analysis set (SAF) included all participants who received at least one dose of rivaroxaban.
Measure: Number; unit: count of participants
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
count of participants
  Major bleeding events | 0 | 0
  Clinically relevant non-major bleeding events | 0 | 0

3. Secondary Outcome: Number of Participants With Symptomatic Recurrent Venous Thromboembolism and Asymptomatic Deterioration in Thrombotic Burden on Repeat Imaging
Description: Symptomatic recurrence of thromboembolism and asymptomatic deterioration was documented using the appropriate imaging test and confirmed by CIAC which was unaware of treatment assignment. Asymptomatic deterioration in thrombotic burden on repeat imaging, as assessed by the CIAC. Adjudication results were the basis for the final analyses.
Time Frame: From start of study drug administration until 30-day post study treatment period
Population: Full analysis set (FAS) included all participants from whom informed consent was obtained and who contributed any data thereafter.
Measure: Number; unit: count of participants
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
count of participants
  Symptomatic recurrent venous thromboembolism | 0 | 0
  Asymptomatic deterioration in thrombotic burden | 0 | 0

4. Primary Outcome: Concentration of Rivaroxaban in Plasma as a Measure of Pharmacokinetics at Day 3
Description: Concentration of pharmacokinetic parameters of rivaroxaban in plasma was evaluated.
Time Frame: 2 to 8 hours post-dose (bid dosing) and 30 minutes to 3 hours post-dose; 7 to 8 hours post-dose on Day 3 (tid dosing)
Population: PKS included all participants with at least one PK sample in accordance with the PK sampling strategy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L)
  30 minutes to 3 hours post-dose: number analyzed (Participants) | 0 | 4
  30 minutes to 3 hours post-dose |  | 32.2879 (267.05)
  2 to 8 hours post-dose: number analyzed (Participants) | 5 | 0
  2 to 8 hours post-dose | 102.3285 (40.36) |
  7 to 8 hours post-dose: number analyzed (Participants) | 0 | 5
  7 to 8 hours post-dose |  | 9.1716 (160.52)

5. Primary Outcome: Concentration of Rivaroxaban in Plasma as a Measure of Pharmacokinetics at Day 8
Description: Concentration of pharmacokinetic parameters of rivaroxaban in plasma was evaluated.
Time Frame: 10 to 16 hours post-dose on Day 8 (bid dosing)
Population: PKS included all participants with at least one PK sample in accordance with the PK sampling strategy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L) | 2.5696 (70.82) | NA (NA) — No participants were analyzed at this time points for tid dosing regimen.

6. Primary Outcome: Change From Baseline in Prothrombin Time at Day 1
Description: Prothrombin time is a global clotting test used for the assessment of the extrinsic pathway of the blood coagulation cascade.
Time Frame: 10-16 hours post-dose on Day 8 (baseline), 2-4 hours after the first dose on Day 1 (bid dosing) and 7-8 hours after the first dose on Day 1 (tid dosing)
Population: Pharmacodynamic (PD) analysis set (PDS) included all participants with at least 1 blood sample for clotting parameters in accordance with the PD sampling strategy were included in the PD analysis.
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
seconds (sec) | 11.6 (17.3) | 0.025 (0.714)

7. Primary Outcome: Change From Baseline in Prothrombin Time at Day 3
Description: as for outcome 6
Time Frame: 10-16 hours post-dose on Day 8 (baseline), 2-8 hours post-dose on Day 3 (bid dosing) and 0.5-3 hours post-dose on Day 3 (tid dosing)
Population: PDS included all participants with at least 1 blood sample for clotting parameters in accordance with the PD sampling strategy were included in the PD analysis.
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
seconds (sec) | 3.74 (2.84) | 1.13 (2.10)

8. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (aPTT) at Day 1
Description: The Activated partial thromboplastin time (aPTT) is a screening test for the intrinsic pathway and is sensitive for deficiencies of factors I, II, V, VIII, IX, X, XI and XII.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
seconds (sec) | 13.6 (12.4) | 2.33 (5.53)

9. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (aPTT) at Day 3
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
seconds (sec) | 7.02 (5.08) | 3.47 (7.59)

10. Primary Outcome: Anti-factor Xa Activity (Anti-Xa) Values at Day 1
Description: The individual anti-Factor Xa activity was determined ex-vivo using a photometric method.
Time Frame: 2-4 hours after the first dose on Day 1 (bid dosing) and 7-8 hours after the first dose on Day 1 (tid dosing)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L) | 63.3 (60.8) | 18.0 (8.37)

11. Primary Outcome: Anti-factor Xa Activity (Anti-Xa) Values at Day 3
Description: The individual anti-Factor Xa activity was determined ex-vivo using a photometric method.
Time Frame: 2-8 hours post-dose on Day 3 (bid dosing) and 0.5-3 hours post-dose on Day 3 (tid dosing)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L) | 67.3 (48.7) | 59.8 (46.8)

12. Primary Outcome: Anti-factor Xa Activity (Anti-Xa) Values at Day 8
Description: The individual anti-Factor Xa activity was determined ex-vivo using a photometric method.
Time Frame: 10-16 hours post-dose on Day 8 (both bid and tid dosing)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
Number analyzed (Participants) | 5 | 5
microgram per liter (mcg/L) | 7.25 (0.00) | 9.92 (5.35)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after the last administration of study drug
Arm/Group | Rivaroxaban (BAY59-7939) Suspension Bid | Rivaroxaban (BAY59-7939) Suspension Tid
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (BAY59-7939) Suspension Bid (N=5) | Rivaroxaban (BAY59-7939) Suspension Tid (N=5)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (BAY59-7939) Suspension Bid (N=5) | Rivaroxaban (BAY59-7939) Suspension Tid (N=5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer shall own the exclusive rights to all results, data, findings, radiological & diagnostic images, discoveries, inventions & specifications, whether patentable or not, that are originated, conceived, derived, produced, discovered, invented or otherwise made by Center, PI and/or Study Team Physicians and/or Members in connection with the performance of the Study (i.e. Results). Contract Partners hereby assign their rights to the Results to Bayer in advance and Bayer accepts such assignment.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02564718/SAP_000.pdf
  • Study Protocol (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02564718/Prot_001.pdf